CLINICAL TRIAL: NCT01514838
Title: A Phase III, Double-Blind, Randomized, Active Controlled, Monotherapy Study to Assess the Efficacy and Safety of ASP1941 in Asian Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Asian Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued due to company's strategic reason
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-2003
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: urine glucose; ipragliflozin; plasma glucose; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glycosuria | interventions — ipragliflozin; Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1941 group (Experimental): Once daily over a 24-week treatment period
  Interventions: Drug: ASP1941; Drug: Placebo
- acarbose group (Active Comparator): Once daily over a 24-week treatment period
  Interventions: Drug: acarbose; Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Other Names: ipragliflozin
  Arms: 1941 group
Drug: acarbose — oral
  Arms: acarbose group
Drug: Placebo — oral, used only during placebo run-in period

SUMMARY:
The purpose of this study is to assess the efficacy of ASP1941 based on the changes in HbA1C as well as its safety in Asian subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a multi-center, active-controlled, double-blind, double-dummy, parallel-group comparative study. After a screening period followed by a placebo run-in period under the single-blind condition, subjects will be randomized to either the ASP1941 or the acarbose group. Subjects will take the study drug under the double-blind condition in the treatment period. After completion of the study drug administration, a follow-up period will be provided.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as type 2 diabetes mellitus patient at least 12 weeks before the study
* stable diet and exercise program for at least 6 weeks before the study
* for the hypoglycemic agent non-naïve subject, subject has been receiving a single hypoglycemic agent or low-dose of a dual combination therapy
* BMI of 20.0 to 45.0 kg/m2
* for the hypoglycemic agent non-naïve subject, subject has a HbA1c value between 6.8 and 10.0% at screening AND has a HbA1c value between 7.0 and 10.0%, inclusive, at run-in period
* for the hypoglycemic agent naïve subject, subject has a HbA1c value between 7.0 and 10.0%, inclusive, at run-in period

Exclusion Criteria:

* type 1 diabetes mellitus
* proliferative diabetic retinopathy
* receiving insulin within 12 weeks prior to the study
* history of clinically significant renal disease(s)
* significant dysuria caused by a neurogenic bladder or a benign prostate hypertrophy etc.
* urinary tract infection or genital infection
* continuous use of systemic corticosteroids, immunosuppressants, or loop diuretics
* history of cerebrovascular attack, unstable angina, myocardial infarction, angioplasty, serious cardiac diseases within 12 weeks prior to the study
* severe infection, serious trauma, or perioperative subject
* known or suspected hypersensitivity to ASP1941, acarbose or other alpha-GI
* history of treatment with ASP1941
* participated in another clinical study, postmarketing study or medical device study within 12 weeks before the study
* serum creatinine value exceeding the upper limit of normal range
* urinary microalbumin/urinary creatinine ratio >300 mg/g

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2012-10-19 (Actual); Study Completion 2012-10-19 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to end of treatment | Baseline and up to 24 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose level | Baseline and up to 24 weeks
Change in fasting serum insulin level | Baseline and up to 24 weeks
Change in body weight | Baseline and up to 24 weeks
Change in body waist circumference | Baseline and up to 24 weeks
Safety assessed by the incidence of adverse events, vital signs safety labo-tests and 12-lead ECG | For 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (15):
- South Korea (8):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Seongnam
  - Seoul
  - Wŏnju
- Taiwan (7):
  - Changha
  - Chiayi City
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=108